CLINICAL TRIAL: NCT00255125
Title: Role of Soy Isoflavones in Prostate Cancer Prevention
Brief Title: Role of Soy Supplementation in Prostate Cancer Development
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLIN-006-05S; NCT00285480 (obsolete NCT alias)
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Prostate Neoplasm
Keywords: Estrogen Receptor; Isoflavones; Prostate Neoplasm; Soy Supplementation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Arm Soy Supplement (Experimental): Soy Supplement
  Interventions: Drug: Soy Supplement

INTERVENTIONS:
Drug: Soy Supplement — Soy protein supplement will be taken for 2-4 weeks until surgery to remove the prostate or start of radiation treatment. Patient will receive 4 capsules twice a day (8 capsules) daily to be taken with water or juice (except grapefruit juice).
  Other Names: Fla-vien
  Arms: Arm Soy Supplement
Drug: Placebo — Placebo will consist of a capsule without the soy protein added to be taken for 2-4 weeks until surgery to remove the prostate or start of radiation treatment. Patient will receive 4 capsules twice a day (8 capsules) daily to be taken with water or juice (except grapefruit juice).
  Other Names: No other name
  Arms: Arm Placebo

SUMMARY:
This is a randomized study evaluating the effectiveness and direct effect a commercial soy supplement has on prostate cancer and normal prostate tissue. Patient will be randomized it either receive placebo or a commercial soy supplement for 2-4 weeks prior to the planned surgery for treatment of their prostate cancer. Patient's blood and prostate tissue will be evaluated to determine the effects of the soy supplement on the prostate tissue.

DETAILED DESCRIPTION:
This is a randomized study evaluating the effectiveness and direct effect a commercial soy supplement has on prostate cancer and normal prostate tissue. Patients will be randomized to either receive placebo or a commercial soy supplement for 2-4 weeks prior to the planned surgery for treatment of their prostate cancer. The specific objectives are:

1. To assess the effect of soy supplementation on endogenous hormone production levels and serum prostate specific antigens.
2. To assess the impact of soy supplementation on estrogen receptor expression(ER).
3. To determine the impact of soy isoflavones on cell cycle regulation and associated gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer.
* Surgical candidate for prostatectomy.
* During study period, must agree not to take new supplements.
* No concurrent chemotherapy, radiation or hormonal therapy.
* No history of prior allergy to soy based products.
* Must not have been taking soy supplements or soy isoflavones within 90 days prior to study enrollment.
* Must be able to safely be on study supplements for period of at least two weeks prior to scheduled prostatectomy.
* Must give written and informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

During study period, must agree not to take new supplements.

* No concurrent chemotherapy, radiation or hormonal therapy.
* No history of prior allergy to soy based products.
* Must not have been taking soy supplements or soy isoflavones within 90 days prior to study enrollment.
* Must be able to safely be on study supplements for period of at least two weeks prior to scheduled

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-09; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vanveldhuizen, MD, Principal Investigator — VA Medical Center, Kansas City MO
Locations (1):
- VA Medical Center, Kansas City MO, Kansas City, Missouri, United States

REFERENCES:
- [Result] Hamilton-Reeves JM, Banerjee S, Banerjee SK, Holzbeierlein JM, Thrasher JB, Kambhampati S, Keighley J, Van Veldhuizen P. Short-term soy isoflavone intervention in patients with localized prostate cancer: a randomized, double-blind, placebo-controlled trial. PLoS One. 2013 Jul 12;8(7):e68331. doi: 10.1371/journal.pone.0068331. Print 2013. PMID 23874588

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm Soy Supplement | Arm Placebo
Started | 42 | 44
Completed | 42 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Prostate cancer patient, randomized between to study groups; all patients with early stage prostate cancer.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm Soy Supplement | Arm Placebo | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (12) | 62 (7) | 62 (12)
Sex/Gender, Customized [Number; unit: participants]
  Male | 42 | 44 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 41 | 42 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 9 | 12
  White | 38 | 31 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 44 | 86

OUTCOME MEASURES:

1. Primary Outcome: Effect of Soy Isoflavones on Serum Testosterone Levels.
Description: Total testosterone (ng/ml) serum levels were measured at the time of enrollment(baseline), after two weeks on soy supplement(time point 1), and just prior to prostatectomy (time point 2). All patients must have completed at least two week of soy supplement or placebo and time point 3 varied depending on date of planned prostatectomy. Results were analyzed and are reported at the two week time period, comparing between patients receiving soy supplement or placebo.
Time Frame: Two weeks
Measure: Mean (80% Confidence Interval); unit: ng/ml
Arm/Group | Arm Soy Supplement | Arm Placebo
Number analyzed (Participants) | 42 | 44
ng/ml | 376 [124 to 528] | 405 [232 to 576]

2. Secondary Outcome: Effect of Soy Isoflavones on Estrogen Receptor Status
Description: Samples of the prostate cancer tissue (paraffin embedded) were sectioned and placed on a glass slide. Using immunohistochemistry and an estrogen receptor antibody, sections were stained and assess to determine the extent of estrogen receptor expression. Patients in the soy supplement arm's samples results were compared to placebo arm results.
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Arm Soy Supplement | Arm Placebo
Number analyzed (Participants) | 42 | 44
pg/mL | 130 (58) | 131 (56)

3. Secondary Outcome: Molecular Effects of Soy Supplementation Compared to Placebo.
Description: Using a tissue microarray targeting the cell cycle, selected fresh prostate cancer samples were evaluated in patients in the soy supplement arm compared to the placebo arm.
Time Frame: One year
Population: Data and project staff no longer available to determine results.
Arm/Group | Arm Placebo | Arm Soy Supplement
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm Soy Supplement | Arm Placebo
Serious Adverse Events (participants affected / at risk) | 2/42 | 6/44
Other Adverse Events (participants affected / at risk) | 9/42 | 4/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm Soy Supplement (N=42) | Arm Placebo (N=44)
Mild gastrointestinal symptoms (Gastrointestinal disorders) | 2 (2) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm Soy Supplement (N=42) | Arm Placebo (N=44)
GI symptoms (Gastrointestinal disorders) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No